CLINICAL TRIAL: NCT01033461
Title: The Effect of the Probiotic L. Paracasei LPC 37 Alone or in Combination With a Calcium Supplement in Healthy Subjects
Brief Title: Combination of Probiotic and Calcium in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H33-08
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Subjects
Keywords: probiotic; lactobacillus paracasei; calcium; faecal microbiota; cholesterol metabolism
MeSH Terms: interventions — Calcium; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- calcium and probiotic (Experimental): intervention
  Interventions: Dietary Supplement: calcium and probiotic
- probiotic (Experimental): intervention
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): placebo, no intervention
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: calcium and probiotic — the subjects consumed for 4 weeks a yoghurt drink enriched with 10e+10 cfu/d L. paracasei LPC 37 and a bread enriched with 1 g pentacalcium phosphate per day
  Arms: calcium and probiotic
Dietary Supplement: probiotic — the subjects consumed a yoghurt drink enriched with 10e+10 cfu/d L. paracasei LPC 37 for 4 weeks
  Arms: probiotic
Other: placebo — the subjects consumed a yoghurt drink without L. paracasei LPC 37 and a bread without pentacalcium phosphate
  Arms: placebo

SUMMARY:
The study was conducted to investigate the effect of the probiotic L. paracasei LPC 37 alone or in combination with a calcium supplement of the human microbiota and further physiological parameters.

DETAILED DESCRIPTION:
Animal studies suggest that calcium beneficially influence the microbiota in the gut. This effect of calcium is due to the formation of amorphous calcium phosphate, which has the ability to bind bile acids and other cytotoxic substances in the gut. The precipitation of the cytotoxic substances leads to a less aggressive environment in the gut and might be stimulate the adhesion of the microbiota.

Thirty-two healthy men and women participated in a placebo-controlled, double-blind and cross over human study. The participants were randomly divided into two groups. All probands consumed a probiotic drink for four weeks (10e+10 CFU/d). Additionally, one group consumed a pentacalcium phosphate-enriched bread (1 g Ca/d) and the other group consumed a bread without pentacalcium phosphate. After a two-week wash-out and a two-week placebo period the invention changed for another four weeks (cross over). At the end of each intervention and placebo period, subjects consumed a defined diet for three days. Furthermore, there was a three-day quantitative stool and urine collection and a fasting venous blood sample was taken.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* blood cholesterol concentration > 5 mmol/l

Exclusion Criteria:

* pregnancy, lactation
* intake of dietary supplements
* intake of prebiotics and probiotics
* chronic diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
faecal microbiota, cholesterol metabolism | 4 weeks

SECONDARY OUTCOMES:
mineral status, immunological parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof.Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutrional Physiology
Locations (1):
- Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutrional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Trautvetter U, Ditscheid B, Kiehntopf M, Jahreis G. A combination of calcium phosphate and probiotics beneficially influences intestinal lactobacilli and cholesterol metabolism in humans. Clin Nutr. 2012 Apr;31(2):230-7. doi: 10.1016/j.clnu.2011.09.013. Epub 2011 Oct 20. PMID 22019281